CLINICAL TRIAL: NCT03139370
Title: A Phase 1 Study Evaluating the Safety and Efficacy of MAGE-A3/A6 T Cell Receptor Engineered T Cells (KITE-718) in HLA-DPB1*04:01 Positive Subjects With Advanced Cancers
Brief Title: Safety and Efficacy of MAGE-A3/A6 T Cell Receptor Engineered T Cells (KITE-718) in HLA-DPB1*04:01 Positive Adults With Advanced Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to the sponsor's decision to discontinue the clinical trial.
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KITE-718-301; 2020-005456-37 (EudraCT Number)
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- KITE-718 (Experimental): Phase 1A: Participants will receive cyclophosphamide and fludarabine conditioning chemotherapy followed by the investigational treatment, KITE-718.
  Phase 1 B: Participants will receive cyclophosphamide and fludarabine conditioning chemotherapy followed by the investigational treatment, KITE-718, at a dose selected based on Phase 1A.
  Interventions: Drug: KITE-718; Drug: Cyclophosphamide; Drug: Fludarabine; Device: MAGE - A3/A6 Screening Test

INTERVENTIONS:
Drug: KITE-718 — A single infusion of autologous genetically modified MAGE-A3/A6 T-cell receptor (TCR) transduced autologous T cells (KITE-718).
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously
Device: MAGE - A3/A6 Screening Test — A screening test for MAGE-A3/A6+ tumors

SUMMARY:
The primary objectives of Phase 1A are to evaluate the safety of KITE-718, determine a recommended Phase 1B dose, and to evaluate the efficacy of KITE-718 in Phase 1B.

DETAILED DESCRIPTION:
Participants found to be human leukocyte antigen (HLA)-DPB1*04:01 positive and whose tumors are MAGE-A3 and/or MAGE-A6 positive can participate if all eligibility criteria are met. Other tests required to determine eligibility include a physical exam, electrocardiogram (ECG) and echocardiogram (ECHO) of the heart, CT or MRI scans, and blood draws. Eligible participants have white blood cells collected by leukapheresis. These cells are genetically modified to make the experimental treatment KITE-718. The desired outcome is that the genetically modified T cells will target tumor cells that express MAGE-A3 and/or MAGE-A6, which are proteins that can be expressed by cancer cells. Participants receive chemotherapy prior to the KITE-718 infusion. After the KITE-718 infusion, participants will be followed for side effects and have scans performed to see any potential impact on their cancers. Study procedures may be performed while hospitalized and/or in the outpatient setting. Subjects who received an infusion of KITE-718 will complete the remainder of the 15 year follow-up assessments in a separate long-term follow-up study, KT-US-982-5968

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years
* Advanced cancer defined as relapsed or refractory disease after a systemic standard of care treatment regimen and, if available, at least one standard of care salvage regimen unless the subject refuses such therapy. Multiple myeloma (MM) subjects must have had both a protease inhibitor (PI) and immunomodulatory drugs (IMiD) as part of the last regimen, or at least 3 prior lines of therapy, including a PI and an IMiD. Additionally, subjects must not have disease amenable to definitive locoregional therapy.
* MAGE-A3/A6 positive tumor as confirmed by the central laboratory
* HLA-DPB1*04:01 positive
* At least 1 measurable lesion on CT or MRI
* No evidence of central nervous system (CNS) disease by MRI or CT of the brain. Note: Prior brain metastasis which have been treated with definitive therapy are eligible provided that the definitive therapy was completed more than six months prior to screening.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Toxicities due to prior therapy must be recovered to baseline or ≤ grade 1, except for clinically non-significant toxicities such as alopecia
* Adequate bone marrow function as evidenced by:

  * Absolute neutrophil count (ANC) ≥ 1000/mm^3
  * Platelet ≥ 100/mm^3
  * Hemoglobin > 8 g/dL
* Adequate renal, hepatic, cardiac, and pulmonary function as evidenced by:

  * Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 cc/min (24-hour urine creatinine clearance is also acceptable)
  * Alanine transaminase (ALT)/aspartate aminotransferase (AST) ≤ 2.5 x upper limit normal (ULN) or ≤ 5 x ULN if documented liver metastases
  * Total bilirubin ≤ 1.5 mg/dL
  * Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an ECHO, and no clinically significant ECG findings (For ejection fraction only, MUGA scan is also acceptable)
  * No clinically significant pleural effusion
  * Baseline oxygen saturation > 92% on room air

Key Exclusion Criteria:

* Malignancy other than non-melanoma skin cancer, carcinoma in situ, or low grade prostate cancer for which watch-and-wait approach is standard of care, unless disease free for at least 3 years
* Clinically significant cardiac disease within last 12 months
* Stroke or transient ischemic attack (TIA) within 12 last months
* Symptomatic deep vein thrombosis or pulmonary embolism within last 6 months, catheter associated thrombosis is not included as exclusion criteria.
* Prior T-cell therapy, including KITE-718 or MAGE-A3/A6-targeting therapy.
* Live vaccine ≤ 4 weeks prior to enrollment
* Systemic corticosteroid therapy within 7 days before enrollment.
* History of severe, immediate hypersensitivity reaction attributed to aminoglycosides
* Presence of fungal, bacterial, viral, or other infection requiring IV antimicrobials for management.
* Presence of any indwelling line or drain. Note: Dedicated central venous access catheters such as a Port-a-Cath or Hickman catheter as well as feeding tubes such as a G-tube, are permitted.
* Primary immunodeficiency
* Autoimmune disease resulting in end-organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years prior to enrollment.
* Known history of infection with HIV, hepatitis B (HBsAg positive), or hepatitis C (anti-HCV positive). A history of treated hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing.
* Females who are pregnant as confirmed by a positive serum or urine pregnancy test or are breastfeeding.
* Individuals of both genders of child-bearing potential who are not willing to practice birth control from the time of consent through 6 months after the completion of KITE-718

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-06-04 (Actual)

PRIMARY OUTCOMES:
Phase 1A - Percentage of Participants Experiencing Adverse Events Defined as Dose-Limiting Toxicities | Up to 21 days
  Dose-limiting toxicity is defined as protocol-defined KITE-718 related events with onset within the first 21 days following KITE-718 infusion.
Phase 1B - Efficacy: Objective Response Rate (ORR) | Up to year 2 for solid tumor participants and up to Year 5 for multiple myeloma participants
  ORR is defined as complete response + partial response for participants evaluated by RECIST v1.1 and very good partial response (VGPR) or better for multiple myeloma participants evaluated by International Myeloma Working Group (IMWG) Consensus Panel 1 Criteria.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to year 2 for solid tumor participants and up to year 5 for multiple myeloma participants
  For participants who experience an objective response, DOR is defined as the time from the date of their first objective response to the date of disease progression per modified RECIST v1.1 or consensus panel 1 criteria or death regardless of cause.
Progression-Free Survival (PFS) | Up to year 2 for solid tumor participants and up to year 5 for multiple myeloma participants
  PFS is defined as the time from the KITE-718 infusion date to the date of disease progression per modified RECIST v1.1 or consensus panel 1 criteria or death from any cause.
Overall Survival | Up to 15 years
  Overall survival is defined as the time from KITE-718 infusion to the date of death.
Percentage of Participants Experiencing Adverse Events | Up to 15 years
Percentage of Participants with Anti-KITE-718 Antibodies | Up to 2 years
Percentage of Participants Experiencing Replication-competent Retrovirus (RCR) | Up to 2 years
Levels of MAGE-A3/A6 TCR-transduced T Cells in Blood | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (12):
- United States (12):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - H. Lee Moffitt Cancer and Research Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Baylor Scott & White Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KITE-718-301